CLINICAL TRIAL: NCT04799769
Title: Clinical Investigation Plan (CIP) for Safety and Performance Study of Large Hole Vascular Closure Device - FRONTIER V Study
Brief Title: Safety and Performance Study of Large Hole Vascular Closure Device - FRONTIER V Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vivasure Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P802-00
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Percutaneous Arteriotomy Closure
Keywords: Arterial Closure; percutaneous arterial closure; large hole arterial closure; large bore arterial closure

STUDY DESIGN:
Intervention Model Description: Prospective, multi-centred, non-randomized study to investigate the safety and performance of the PerQseal® +
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Device (Experimental): Investigational Device Arm
  Interventions: Device: Percutaneous arterial closure device

INTERVENTIONS:
Device: Percutaneous arterial closure device — Large hole percutaneous arterial closure device

SUMMARY:
This study will be a prospective, multi-centred, non-randomized study to investigate the safety and performance of the PerQseal® + in up to 90 patients in up to 8 European investigational sites. The PerQseal® + shall be indicated for the percutaneous closure of femoral artery punctures and to induce arterial haemostasis in patients undergoing endovascular procedures requiring an arteriotomy created with 14 - 22F sheaths (arteriotomy up to 26 F).

DETAILED DESCRIPTION:
The study will be designed to be a phased study with an initial enrolment of 25 subjects in phase 1. An interim analysis may be performed after phase 1 and the remainder (up to 65 subjects) may be enrolled as part of phase 2.

The study shall not be blinded prior to, during or post the procedure. All patients undergoing an endovascular procedure requiring an arteriotomy created by 14 to 22 F sheaths, via the common femoral artery will be screened against the inclusion/exclusion criteria. If the patient meets the requirements of the clinical investigation, they shall be invited to participate, provide informed consent and shall subsequently be assigned a 'Subject Number'. The closure will be percutaneous. An optional adjunctive endovascular balloon may be used to control bleeding. All safety data from the study will be assessed by the Data Safety Monitoring Committee on a continuous basis.

The Purpose of the Study is to assess safety and performance of the PerQseal® + Closure Device when used with the L PerQseal® Introducer to percutaneously close femoral artery punctures and to induce arterial haemostasis in patients undergoing endovascular procedures requiring an arteriotomy created by 14 to 22 F sheaths.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Subject is willing and able to provide appropriate study-specific informed consent, follow protocol procedures, and comply with follow-up visit requirements.
* Clinically indicated for an endovascular procedure using a common femoral arteriotomy created by a 14 - 22 F sheath.

General Exclusion Criteria:

* Severe acute non-cardiac systemic disease or terminal illness with a life expectancy of less than four months.
* Evidence of systemic bacterial or cutaneous infection, including groin infection.
* Known bleeding diathesis (including sever liver disease), definite or potential coagulopathy, platelet count < 100,000/µl or patients on long term anticoagulants with an INR greater than 2 at time of procedure or known type II heparin-induced thrombocytopenia.
* Previous groin surgery within the region of the ipsilateral access.
* Severe; claudication or peripheral vascular disease (e.g. Rutherford category 3 or greater or ABI < 0.5), documented untreated iliac artery diameter stenosis > 50% or previous bypass surgery/stent placement in the common femoral artery of ipsilateral limb.
* Known allergy to any of the materials used in the PerQseal® + or PerQseal® Introducer (refer to Investigator's Brochure for materials list).
* Subject has undergone a percutaneous procedure using a non-absorbable vascular closure device (excluding suture mediated) for haemostasis in the ipsilateral target leg.
* Patients that have undergone a percutaneous procedure in the ipsilateral leg, within the previous 30 days.
* Patients that have undergone a percutaneous procedure using an absorbable intravascular closure device for haemostasis, in the ipsilateral leg, within the previous 90 days.
* Evidence of arterial diameter stenosis > 20% or anterior or circumferential calcification within 20 mm proximal or distal to target arteriotomy site based on pre-procedure CT angiography.
* Females who are pregnant or lactating or in fertile period not taking adequate contraceptives. A pregnancy test may be performed.
* Patients that have a lower extremity amputation from the ipsilateral or contralateral limb.
* Target puncture site is located in a vascular graft.

Procedural Exclusion Criteria:

* Arterial access other than common femoral artery obtained for ipsilateral target leg.
* Subject has a tissue tract expected to be greater than 10 cm.
* Significant blood loss/transfusion (defined as requiring transfusion of 4 or more units of blood products) during index procedure or within 30 days prior to index procedure.
* Unstable blood pressure or heart rate, symptoms of shock or systolic blood pressure greater than 160 mmHg (maybe controlled by pacing or pharmacologically eg. vasodilator such as nitrates etc.).
* Activated clotting time (ACT) > 350 seconds immediately prior to sheath removal or if ACT measurements are expected to be > 350 seconds for more than 24 hours after index procedure.
* Target arteriotomy is in the profunda femoris or superficial femoral artery or is in common femoral artery, but within 15 mm proximal of the bifurcation of the Superficial Femoral /Profunda Femoris artery.
* PerQseal® Introducer-sheath to ipsilateral femoral artery diameter ratio is greater than or equal to 1.05. (vessel lumen diameter of less than 7 mm.)
* Subjects with an acute haematoma of any size, arteriovenous fistula or pseudoaneurysm at the target access site; or any evidence of arterial laceration or dissection within the external iliac or femoral artery before the use of the PerQseal® + Closure Device.
* Use of thrombolytic agents within 24 hours prior to or during the endovascular procedure which causes fibrinogen < 100 mg/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-01-10 (Estimated); Study Completion 2023-03-10 (Estimated)

PRIMARY OUTCOMES:
Primary Safety | 1-month post implantation (inclusive)
  Major vascular access site complication rate related to the PerQseal® + Closure Device

SECONDARY OUTCOMES:
Secondary Safety | 1-month post implantation (inclusive)
  Minor vascular access site complication rate related to the PerQseal® + Closure Device
Performance | Up to 5 days post implantation
  Technical success rate for the PerQseal® + Closure Device

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (4):
  - SHG-Kliniken Völklingen, Völklingen, Saarland
  - Leipzig University Hospital, Leipzig, Saxony
  - University Hospital Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - St. Franziskus-Hospital, Münster, Westphalia
- Erasmus Hospital, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No